CLINICAL TRIAL: NCT04326738
Title: The Effect of Midazolam on Dexamethasone-induced Perineal Pruritus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Ma Hong, Affiliated Hosptial of Yangzhou University, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-YKL-003
Record Dates: First submitted 2020-03-26; First posted 2020-03-30 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Pruritus
Keywords: midazolam; Dexamethasone; pruritus
MeSH Terms: conditions — Pruritus | interventions — Midazolam; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal saline (N) group (Placebo Comparator): N group received corresponding intravenous normal saline of 1ml·kg-1.
  Interventions: Drug: normal saline
- midazolam (M) group (Active Comparator): M group received intravenous injection of 0.03mg·kg-1 (1mg·ml-1) midazolam.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — M group received intravenous injection of 0.03mg·kg-1 (1mg·ml-1) midazolam, After 1 min, both groups received intravenous injection of dexamethasone sodium phosphate injection of 10mg (injection was completed in 2s)
  Arms: midazolam (M) group
Drug: normal saline — N group received corresponding intravenous normal saline of1ml·kg-1 .
  Arms: normal saline (N) group

SUMMARY:
Dexamethasone is commonly used in clinical practice.However, intravenous dexamethasone sodium phosphate may cause perineal discomfort.With the popularization of comfortable medical technology, patients have higher and higher requirements for comfortable medical treatment.Perineal pruritus caused by intravenous dexamethasone sodium phosphate may cause adverse physiological and psychological effects on patients and increase the incidence of unpleasant experiences during anesthesia.Therefore, it is very important to find a practical and effective method of inhibition.Midazolam is a water-soluble benzodiazepine commonly used in clinical practice, which has been proved to effectively inhibit the itching caused , while its effect on the itching caused by dexamethasone has not been reported.By observing the effect of pre-injection midazolam on the perineal itching caused by dexamethasone sodium phosphate, this experiment intends to preliminarily explore its possible mechanism .

DETAILED DESCRIPTION:
Nighty patients scheduled for selective surgery,aged 18-65years,ASA physical status I~II,BMI 18~30kg·m-2 were selected in this study.The patients were equally randomized into two groups: midazolam (M) group and normal saline (N) group, 45 cases in each group. Before anesthesia induction, M group received intravenous injection of 0.03mg·kg-1 (1mg·ml-1) midazolam, while N group received corresponding intravenous normal saline of the same volume. After 1 min, both groups received intravenous injection of dexamethasone sodium phosphate injection of 10mg (injection was completed in 2s). The anesthesiologist assessed perineal irritation in both groups and recorded the number of cases,visual analogue scores (VAS) ,duration of itching or pain,Ramsay scores and observed the occurrence of adverse reactions such as dizziness and respiratory depression in the two groups.

ELIGIBILITY:
Inclusion Criteria:

the undergoing elective surgery patients, ages 18 to 65 years, ASA Ⅰ or Ⅱ level, body mass index (BMI) of 18 ~ 30 kg · m-2.

Exclusion Criteria:

diabetes mellitus, paresthesia, allergy to narcotic drugs, routine preoperative use of narcotic analgesics, long-term use of hormones, drug and alcohol abuse, communication disorders in psychiatric disorders, pregnancy or lactation, and patients with severe systemic diseases and unwilling to undergo the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
itching measured by visual analogue scores | in 3 minutes
  visual analogue scores(VAS)VAS 0 means no discomfort, 1-3 as mild, 4-6 as moderate, and 7-10 as severe

SECONDARY OUTCOMES:
Ramsay scores | in 3 minutes
  1 point, not quiet; 2 points, quiet cooperation; 3, drowsiness, ability to follow instructions; 4 points, sleep state, can wake up; 5 points, slow response; 6 points, deep sleep state
the occurrence of adverse reactions | in 3 minutes
  dizziness and respiratory depression

CONTACTS AND LOCATIONS:
Overall Officials: mei yu liu, Study Director — Yangzhou University
Locations (1):
- Affiliated hospital of yangzhou university, Yangzhou, Jiangsu, China